CLINICAL TRIAL: NCT06651489
Title: Efficacy of Guselkumab in the Treatment of Hailey Hailey Disease: An Open-label, Proof of Concept Study
Brief Title: Efficacy of Guselkumab in Treating Hailey Hailey Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000038224
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Hailey Hailey Disease
MeSH Terms: conditions — Pemphigus, Benign Familial | interventions — guselkumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Guselkumab (Experimental): Participants with HHD with be given guselkumab
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Subcutaneous injection of 100 mg at Weeks 0, 4, 12, and 20
  Other Names: Tremfya

SUMMARY:
Hailey-Hailey disease (HHD) is a debilitating genetic skin disorder, affecting mainly body folds with erythema and painful erosions and blisters. Histopathological findings include epidermal hyperplasia, suprabasilar clefting, dyskeratosis and acantholysis of keratinocytes. A final diagnosis of HHD is usually confirmed based on clinical and histopathological findings in line with genetic testing.

Several treatment options have been proposed for this chronic and disabling disorder, however, there is no reproducibly effective therapeutic for it.

The primary objective is to evaluate the treatment response of guselkumab. Single-center, non-randomized, single-arm, open-label, phase II trial to evaluate the efficacy and safety of guselkumab for the treatment of patients with HHD.

DETAILED DESCRIPTION:
Several treatment options have been proposed for HHD as chronic and disabling disorder, however, there is no reproducibly effective therapeutic for it.

The primary objective is to evaluate the treatment response of guselkumab. After the participant has been deemed an appropriate candidate for the study and has signed the consent form, they will be enrolled. All participants will be started on guselkumab 100mg at the FDA-approved psoriasis dose and will be seen for clinical follow-up 4, 12, 24 weeks after initiation of therapy. A 12-week follow-up period will be conducted post-administration of the final dose of guselkumab to monitor safety. Laboratory monitoring including Complete Blood Count, Basic metabolic panel, Liver function tests, and pregnancy test (if applicable) will also be performed at 1 month, 3 months, and 6 months after starting therapy. At each visit except Week 20 a full H&P, complete Review of Systems and physical examination will be performed. Outcomes will be assessed and full-body photography will be performed at each visit except Week 20. Research tissue samples (skin biopsies) will be obtained at baseline (prior to therapy) after 24 weeks of treatment in all participants. Research blood will be obtained at screening, baseline and after 4, 12, and 24 weeks of guselkumab therapy.

ELIGIBILITY:
Inclusion Criteria:

* A documented diagnosis of Hailey-Hailey disease confirmed with clinical, and histopathologic findings
* Disease affecting more than one body site with at least moderate severity
* If patients are taking other systemic therapies for their HHD (antibiotics, prednisone), they must be taking a stable dose of the other medication(s) for at least 3 months with no plans to change the regimen in the next 6 months. With the exception of antibiotics, methotrexate or low dose prednisone (less than 5 mg daily), use of concomitant immunosuppressants, e.g. azathioprine, etc. and biologics other than TNF-α inhibitors will not be permitted.
* Patients must be willing to have skin biopsies, blood collection, and total body photography and to comply with clinic visits

Exclusion Criteria:

* Patients with a history of malignancy (except history of successfully treated basal cell or squamous cell carcinoma of the skin over six months prior to first study drug administration).
* Patients known to be HIV or hepatitis B or C positive.
* Patients planning to receive live vaccines during the duration of the study.
* Patients with a positive tuberculin skin test or positive QuantiFERON TB test.
* Patients with significant hepatic impairment (Child-Pugh class B and C).
* Patients taking immunosuppressive and biologic medications, except for methotrexate, low-dose prednisone, and TNF-α inhibitors, including but not limited to mycophenolate mofetil, azathioprine, tacrolimus, and cyclosporine.
* Are pregnant, nursing, or planning a pregnancy while enrolled in the study or for 12 weeks after the study agent injection for women or are planning to father a child while enrolled in the study or for 12 weeks after the last study agent injection.
* Prior biologic use within the last 3 months.
* Participant has known allergies, hypersensitivity, or intolerance to guselkumab or its excipients (refer to Investigator's brochure)
* Presence of significant uncontrolled respiratory, hepatic, renal, endocrine, hematologic, neurologic, or neuropsychiatric disorders, or abnormal laboratory screening values that, in the opinion of the investigator, pose an unacceptable risk to the subject if participating in the study or of interfering with the interpretation of the data.
* Active, untreated, acute infection, or immunocompromised to an extent that participation in the study would pose an unacceptable risk to the subject based on the investigator's clinical assessment.
* Symptomatic herpes zoster infection within 12 weeks of screening or recurrent or disseminated (even a single episode) herpes zoster.
* Symptomatic herpes simplex or disseminated (even a single episode) herpes simplex at the Week 0 (baseline) visit.
* Patients with the potential for keloid formation, e.g. patients with a propensity for keloid formation, defined as a personal history of 3 or more keloids.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Physician's Global Assessment (PGA) score | baseline and week 24
  The PGA is a widely recognized and frequently utilized scale for evaluating treatment outcomes in clinical trials, spanning across both adult and pediatric populations. It is a straightforward tool with easily interpretable results. . In order to conduct this assessment, a healthcare provider or physician relies on a comprehensive analysis of data gathered from all aspects of the patient's medical history and condition. Scoring is based on a 9 point Likert scale ranging from Markedly Improved (+4) to Markedly Worse (-4).
Change in Ichthyosis Scoring System (ISS) score | baseline and week 24
  ISS is a reliable system to measure global ichthyosis severity in adults and children. The body is divided into 10 regions, and Likert scales (0-4) are used to quantify scale and erythema, with extensive descriptors and photographic standards. The ISS score takes values from 0 to 75. Higher scores indicate more severe injury.

SECONDARY OUTCOMES:
Change in Dermatology Life Quality Index (DLQI) score | week12 and week 24
  The Dermatology Life Quality Index (DLQI) is a questionnaire consisting of ten questions used to gauge how a skin disease affects an individual's quality of life. Each question evaluates the influence of the skin condition on the patient's life during the preceding week. Each question is rated on a scale from 0 to 3, resulting in a potential score range from 0 (indicating no impact of the skin disease on quality of life) to 30 (representing the maximum impact on quality of life). A decrease in DLQI scores indicates improved well-being.
Changes in Health-Related Quality of Life (HRQoL) score | baseline, week12 and week 24
  HRQoL is an evaluation of how an individual's overall well-being could be influenced over a period of time due to a medical condition, disability, or disorder. The scale comprises three components. The first module which will be used in this study, known as the Core Healthy Days module, includes a single item prompting respondents to assess their overall health using a 5-point scale (1 = excellent; 3 = good; 5 = poor). Within this module, there are also three additional items that inquire about the number of days when respondents experienced poor physical health, poor mental health, and days when their health disrupted their daily activities. To calculate an unhealthy day's score, researchers sum the number of days marked as physically unhealthy and mentally unhealthy. The highest possible score is 30 unhealthy days. Lowest score is 0 unhealthy days.
Physician's Global Assessment (PGA) scores | baseline and weeks 4,12 and 24.
  Physicians evaluate the overall severity of ichthyosis based on clinical judgment, considering factors such as scaling, erythema, and patient-reported symptoms. Scoring is based on a 9 point Likert scale ranging from Markedly Improved (+4) to Markedly Worse (-4). Improvement in PGA involves a decrease in overall severity as judged by the physician.
Changes in cytokines | baseline and weeks 4,12 and 24
  Cytokine levels (pg/ml) will be assessed in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Keith Choate, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Church Street Research Unit, Yale Center for Clinical Investigation, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No